CLINICAL TRIAL: NCT05088837
Title: Effect of Muscle Energy Technique on Postpartum Sacroiliac Joint Dysfunction
Brief Title: Muscle Energy Technique on Sacroiliac Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cairo Un113
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Sacroiliac Disorder
Keywords: Muscle energy technique; sacroiliac dysfunction; ice and heat pack
MeSH Terms: interventions — Ice

STUDY DESIGN:
Intervention Model Description: Group (A) (Control group): consisted of 20 patients, they received muscle energy technique for 12 sessions, 3 sessions / week. Group (B) (Study group): consisted of 20 patients, they received alternative heat and ice for another 20 minutes /session (10 minutes for each).
Who Masked: Outcomes Assessor
Masking Description: An independent individual randomly appointed to all participants to either group (A) (n=20) or group (B) (n=20) by numbers that were picked from the closed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- muscle energy technique (Experimental): muscle energy technique was performed in the form of post-isometric relaxation technique for iliopsoas, hamstrings, and erector spinae and quadratus lumborum muscles, it was done 3 times per session for 12 sessions.
  Interventions: Other: muscle energy technique
- ice and heat packs (Experimental): Alternating ice and heat (20 min , 10 heat,10 cold),3times per week for 12sessions.
  Interventions: Other: ice and heat packs

INTERVENTIONS:
Other: muscle energy technique — MET was performed in the form of post-isometric relaxation technique for iliopsoas, hamstrings, and erector spinae and quadratus lumborum muscles. the limb was taken very slightly beyond the restriction barrier and was held there for 10-30 seconds, it was done 3 times per session for 12 sessions.
  Arms: muscle energy technique
Other: ice and heat packs — Applying 20 minutes: 10 minutes hot,10 minutes cold on sacroiliac area, 3 times per week for 12 sessions
  Arms: ice and heat packs

SUMMARY:
Sacroiliac pain is a huge problem in women during pregnancy and postpartum period. Muscle energy technique has potential effect in decreasing the pain and disability

DETAILED DESCRIPTION:
A sample of forty women diagnosed with postpartum sacroiliac dysfunction, their ages ranged from 20 to 40 years and their BMI was ranged from 25-30 kg / m2 participated in this study, they were selected and divided randomly into 2 equal groups (A&B). Group (A) (Control group): consisted of 20 patients, they received muscle energy technique for 12 sessions, 3 sessions / week. Group (B) (Study group): consisted of 20 patients, they received alternative heat and ice for another 20 minutes /session (10 minutes for each). All patients in both group were evaluated at the beginning of the study and after 12 sessions through measuring pain intensity using visual analog scale and disability using oswestry disability index (ODI)

ELIGIBILITY:
Inclusion Criteria:

* Their ages ranged from 20 to 40 years .
* Their BMI was ranged from 25-30 kg / m2

Exclusion Criteria:

* hip fracture,
* SIJ infection.
* scoliosis

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale Visual anlage scale | 4 weeks
  It was used for determining pain intensity before and after the treatment course for each patients in both groups (A&B). Visual analogue scale is a-10 centimeters line, at one end was written (no pain = zero) and at the other end was written (worst pain the patient ever felt = 10)

SECONDARY OUTCOMES:
Oswestry disability index | 4 weeks
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, were used to measure the level of disability before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ghada Ebrahim Elrefaye, Giza, Egypt